CLINICAL TRIAL: NCT05257239
Title: Acceptability and User Perceptions of Artificial Intelligence-based Mobile Applications
Brief Title: Acceptability and User Perceptions of Artificial Intelligence-based Mobile Applications Adoption for Weight Management: A Sequential Explanatory Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jocelyn Chew, Research Fellow, National University Health System, Singapore
Other Study IDs: 2021/00834
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Weight Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — National University Health System,
  Other Names: National University Health System,

SUMMARY:
To understand the user perceptions of AI and non-AI-based mobile apps for weight management in people with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited if they are above 21 years old, have a BMI ≥23kg/m2 and understand English language.

Exclusion Criteria:

* There will be no exclusion criteria to maximize representation of the general population of Singaporean who are overweight and obese.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Singaporean population
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-02-17 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Unified Theory of Acceptance and Use of Technology 2 (UTAUT2) | 2021-2023

SECONDARY OUTCOMES:
Qualitative interviews | 2021-2023

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No